CLINICAL TRIAL: NCT01063868
Title: A One-Year, Randomized, Open-Label, Parallel-Group, Multiple-Dose Long-Term Safety Study With Controlled Adjustment of Dose of Tapentadol Extended-Release (ER) and Oxycodone Controlled-Release (CR) in Subjects With Chronic, Painful Diabetic Peripheral Neuropathy (DPN)
Brief Title: A Long-term Safety Study With Tapentadol ER and Oxycodone CR in Patients With Moderate to Severe Pain Due to Chronic, Painful Diabetic Peripheral Neuropathy (DPN)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016978; R331333PAI3028 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); KF57 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuropathy, Painful; Diabetic Polyneuropathy
Keywords: Diabetic neuropathy; Painful; Polyneuropathy; Peripheral neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Polyneuropathies; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Tapentadol extended release (ER) 100 150 200 250 mg twice daily for 52 weeks
  Interventions: Drug: Tapentadol extended release (ER)
- 002 (Active Comparator): Oxycodone controlled release (CR) 20 30 40 50 mg twice daily for 52 weeks
  Interventions: Drug: Oxycodone controlled release (CR)

INTERVENTIONS:
Drug: Tapentadol extended release (ER) — 100, 150, 200, 250 mg twice daily for 52 weeks
  Arms: 001
Drug: Oxycodone controlled release (CR) — 20, 30, 40, 50 mg twice daily for 52 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety profile of orally administered tapentadol ER dosages of 100 to 250 mg twice daily in patients with chronic, painful diabetic peripheral neuropathy (DPN) over long-term exposure of up to 1 year.

DETAILED DESCRIPTION:
This is a randomized, open-label, active-controlled, multicenter study evaluating the safety profile of orally administered tapentadol, using the extended release tamper-resistant formulation (TRF), at dosages of 100 to 250 mg twice daily in patients with moderate to severe pain due to chronic, painful DPN. The study consists of 1) a 13-day screening period, a 3-7-day washout period (where patients are to stop taking their pain medication), a 1-day pretitration pain-intensity evaluation period (where patients will record their 24-hour pain intensity), and a 3-week, open-label titration period (patients will receive either tapentadol ER or oxycodone CR study drug in a 3 to 1 ratio), 2) a 49-week, open-label maintenance phase, and 3) a posttreatment phase of approximately 10 to 14 days. The study will evaluate the safety and tolerability of orally administered tapentadol ER by vital signs, physical examinations, clinical laboratory tests, 12-lead electrocardiograms (ECGs), opioid withdrawal scales, assessment of patient-reported constipation, standardized neurologic examinations and monitoring of adverse events. Assessments of pain relief include the pain intensity numerical rating scale, and patient global impression of change scale (PGIC). The total duration of study drug treatment for each patient will be approximately 52 weeks. Titrate tapentadol ER 50 mg twice daily or oxycodone CR 10 mg twice daily to patient's optimal dose ranging between 100 mg and 250 mg twice daily or 20 and 50 mg twice daily, respectively. All doses of study medication will be taken orally with or without food for a maximum timeframe of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years or older
* Patients with Type 1 or 2 diabetes mellitus must have a documented clinical diagnosis of painful diabetic peripheral neuropathy with symptoms and signs for at least 6 months, and pain present at the time of screening
* Diagnosis must include pain plus reduction or absence of pin sensibility and/or vibration sensibility on Total Neuropathy Score - Nurse (TNSn) examination in lower and/or upper extremities at screening
* The investigator considers the patient's blood glucose to be controlled by diet, or hypoglycemics, or insulin for at least 3 months prior to enrolling in the study (this control should be documented by figures of glycated hemoglobin (HbA1c) no greater than 11% at screening)
* Patients have been taking analgesic medications for the condition for at least 3 months prior to screening (patients taking opioid analgesics must be dissatisfied with current treatment, and patients taking non-opioid analgesics must be dissatisfied with current analgesia)
* Patients currently requiring opioid treatment must be taking daily doses of an opioid-based analgesic equivalent to <=160mg of oral morphine
* Patients with baseline score for average pain intensity in the previous 24 hours of =>4 on the 11-point numerical rating scale (NRS) at the beginning of the titration period

Exclusion Criteria:

* Significant pulmonary, gastrointestinal, endocrine, metabolic (except diabetes mellitus), neurological, psychiatric disorders (resulting in disorientation, memory impairment or inability to report accurately as in schizophrenia, Alzheimer's disease)
* History of moderate to severe hepatic impairment
* Severely impaired renal function
* Clinically significant laboratory abnormalities
* Clinically significant cardiac disease
* History of seizure disorder or epilepsy
* History of any other clinically significant disease that in the investigator's opinion may affect efficacy or safety assessments or may compromise patient safety during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (23):
- United States (23):
  - Mesa, Arizona
  - Tucson, Arizona
  - Fruitland Park, Florida
  - New Port Richey, Florida
  - Oviedo, Florida
  - Tampa, Florida
  - Libertyville, Illinois
  - Franklin, Indiana
  - Paducah, Kentucky
  - Wellesley Hills, Massachusetts
  - Albuquerque, New Mexico
  - New York, New York
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Tulsa, Oklahoma
  - Greer, South Carolina
  - Dallas, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Tapentadol ER: Tapentadol extended release (ER) 100 150 200 250 mg twice daily for 52 weeks
- Oxycodone CR: Oxycodone controlled release (CR) 20 30 40 50 mg twice daily for 52 weeks
Period: Overall Study
Arm/Group | Tapentadol ER | Oxycodone CR
Started | 35 | 12
Completed | 0 | 0
Not Completed | 35 | 12
Not completed — Adverse Event | 9 | 7
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Study Terminated By Sponsor | 23 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol ER | Oxycodone CR | Total
Number analyzed (Participants) | 35 | 12 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 9 | 35
  >=65 years | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.41) | 60.1 (9.23) | 58.2 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 2 | 17
  Male | 20 | 10 | 30
Region Enroll (United States of America) [Number; unit: participants] | 35 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAE)
Description: The number of participants who reported a TEAE during the treatment period. TEAE was defined as any adverse event that started or worsened on or after the start of the study medication and up to 3 days after the discontinuation of the study medication.
Time Frame: Entire Study
Population: Safety analysis set (All randomized participants who took at least one dose of study medication).
Measure: Number; unit: participants
Arm/Group | Tapentadol ER | Oxycodone CR
Number analyzed (Participants) | 35 | 12
participants | 23 | 11

ADVERSE EVENTS:
Description: Only participants who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total number of participants with Non-Serious Adverse Events.
Arm/Group | Tapentadol ER | Oxycodone CR
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/12
Other Adverse Events (participants affected / at risk) | 19/35 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol ER (N=35) | Oxycodone CR (N=12)
Nausea (Gastrointestinal disorders) | 7 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Somnolence (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Asthenia (General disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Early termination, due to sponsor's discretion, lead to only 47 patients out of the 800 planned (5.9%) being available for analysis. The data should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less